CLINICAL TRIAL: NCT01305928
Title: Increasing Post-Discharged Follow-Up Among Hospitalized Smokers
Brief Title: Hospitalized Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Kimber Richter, PhD, MPH, MA, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2011-02-24; First posted 2011-03-01 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Hospitalized Smokers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fax (Active Comparator)
  Interventions: Other: Fax
- Warm Hand-off (Experimental)
  Interventions: Other: Warm Hand-off

INTERVENTIONS:
Other: Warm Hand-off — Warm Hand-Off
  Staff brief intervention and warm hand-off (5 min):
  * Assess withdrawal, need for medication change
  * Describe warm hand-off process
  * Provide 2-page flyer
  * Perform call, leave room
  * Notify patients' nurse patient is talking to quitline
  Quitline session (20 min):
  * Collect minimum data set
  * Explore thoughts/feelings toward quitting
  * Provide medication education
  * Build plan to stay quit
  * Schedule next call
  Staff check-back (5 min):
  * Ask patient how session went
  * Ask if patient requests cessation medication script on discharge
  Arms: Warm Hand-off
Other: Fax — Fax
  Staff standard in-patient session: (30 minutes):
  * Assess withdrawal, need for medication change
  * Conduct assessment of smoking history, interest in quitting
  * Explore relevance, risks, rewards, and roadblocks (4Rs) related to smoking and quitting
  * Provide 2-page flyer
  * Provide medication education
  * Build plan to stay quit
  * Describe fax-referral process
  * Ask if patient requests cessation medication script on discharge
  Arms: Fax

SUMMARY:
Post-discharge support is a key component of effective treatment for hospitalized smokers, but very few hospitals provide it. Linking hospitalized smokers with free, proactive tobacco quitlines is an ideal way to provide supportive contact at discharge, because quitlines are effective and cost effective for smoking cessation. Many hospitals are beginning to fax-refer smokers to quitlines at discharge. Fax referral is convenient and is part of the current culture of medical communication channels. However, less than half of fax-referred smokers are successfully contacted and enrolled in quitline services. "Warm hand-off" is a novel approach to care transitions in which health care providers directly link patients that have substance abuse and mental health problems with specialists, using face-to-face or phone transfer. Warm hand-off achieves very high rates of treatment enrollment for these highly vulnerable groups.

DETAILED DESCRIPTION:
The objective if this application is to determine the relative effectiveness, and cost-effectiveness, of warm hand-off versus fax referral for linking hospitalized smokers with tobacco quitlines. This study employs a two-arm, individually randomized design. It is set in two large Kansas hospitals that have dedicated tobacco treatment interventionists on staff.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include being residents of Kansas,
* aged 18 years and older,
* have smoked at least 1 cigarette in the 30 days prior to admission,
* speak Spanish or English,
* and wish to remain abstinent after they are discharged
* Patients who are discharged to another facility (for long term care or rehabilitation) will be included in the trial.

Exclusion Criteria:

* Exclusion criteria include lacking access to a telephone post-discharge,
* acute life-threatening medical conditions (for example, cardiac arrest, acute respiratory failure, septic shock),
* communication barriers (intubation, unable to speak or hear),
* altered mental status,
* severe unstable psychiatric disorder (acute psychosis),
* terminal illness with less than a 12 month life expectancy
* non-Kansans because residents of other states may receive quitline services from a different vendor which would confound intervention effects and make it difficult to obtain quitline adherence data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1054 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence, verified smoking cessation | up to 6 months
  To test the effects of warm hand-off versus fax referral on smoking cessation

SECONDARY OUTCOMES:
Enrollment in quitline services and adherence to quitline counseling sessions | up to 6 months
  To test the effects of warm hand-off versus fax referral on enrollment and adherence in quitline services
To examine the costs to providers and participants of the intervention and control conditions | up to 6 months
  To examine the cost-effectiveness of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kimber Richter, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Triant VA, Grossman E, Rigotti NA, Ramachandran R, Regan S, Sherman SE, Richter KP, Tindle HA, Harrington KF. Impact of Smoking Cessation Interventions Initiated During Hospitalization Among HIV-Infected Smokers. Nicotine Tob Res. 2020 Jun 12;22(7):1170-1177. doi: 10.1093/ntr/ntz168. PMID 31687769
- [Derived] Mussulman LM, Scheuermann TS, Faseru B, Nazir N, Richter KP. Rapid relapse to smoking following hospital discharge. Prev Med Rep. 2019 May 23;15:100891. doi: 10.1016/j.pmedr.2019.100891. eCollection 2019 Sep. PMID 31193919
- [Derived] Liebmann EP, Scheuermann TS, Faseru B, Richter KP. Critical steps in the path to using cessation pharmacotherapy following hospital-initiated tobacco treatment. BMC Health Serv Res. 2019 Apr 24;19(1):246. doi: 10.1186/s12913-019-4059-4. PMID 31018852
- [Derived] Scheuermann TS, Preacher KJ, Carlini BH, Bush T, Magnusson B, Nazir N, Richter KP. Predictors of engagement in post-discharge quitline counseling among hospitalized smokers. J Behav Med. 2019 Feb;42(1):139-149. doi: 10.1007/s10865-018-9951-6. Epub 2018 Jul 19. PMID 30027388
- [Derived] Mussulman LM, Faseru B, Fitzgerald S, Nazir N, Patel V, Richter KP. A randomized, controlled pilot study of warm handoff versus fax referral for hospital-initiated smoking cessation among people living with HIV/AIDS. Addict Behav. 2018 Mar;78:205-208. doi: 10.1016/j.addbeh.2017.11.035. Epub 2017 Nov 26. PMID 29216569
- [Derived] Richter KP, Faseru B, Shireman TI, Mussulman LM, Nazir N, Bush T, Scheuermann TS, Preacher KJ, Carlini BH, Magnusson B, Ellerbeck EF, Cramer C, Cook DJ, Martell MJ. Warm Handoff Versus Fax Referral for Linking Hospitalized Smokers to Quitlines. Am J Prev Med. 2016 Oct;51(4):587-96. doi: 10.1016/j.amepre.2016.04.006. PMID 27647059
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Richter KP, Faseru B, Mussulman LM, Ellerbeck EF, Shireman TI, Hunt JJ, Carlini BH, Preacher KJ, Ayars CL, Cook DJ. Using "warm handoffs" to link hospitalized smokers with tobacco treatment after discharge: study protocol of a randomized controlled trial. Trials. 2012 Aug 1;13:127. doi: 10.1186/1745-6215-13-127. PMID 22853047